CLINICAL TRIAL: NCT05212337
Title: Effect of a Single-dose Denosumab on Semen Quality in Infertile Men (FITMI): A Randomized Controlled Trial
Brief Title: FITMI - First In Treating Male Infertility
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Martin Blomberg Jensen (Other)
Responsible Party: Sponsor-Investigator, Martin Blomberg Jensen, Medical Doctor, Rigshospitalet, Denmark
Organization: Rigshospitalet, Denmark (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 19642021
Record Dates: First submitted 2022-01-03; First posted 2022-01-28 (Actual); Last update posted 2024-11-15 (Actual); Status verified 2024-11

CONDITIONS: Infertility, Male
MeSH Terms: conditions — Infertility, Male | interventions — Denosumab; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: Interim analysis will be forward to study committee to evaluate data and decide whether study should proceed to be stopped
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: groups designated with X and Y
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Denosumab (Active Comparator): Subcutaneous injection with 60 mg Denosumab once
  Interventions: Drug: Denosumab
- Placebo (Placebo Comparator): Subcutaneous injection with NaCl once
  Interventions: Drug: Sodium chloride

INTERVENTIONS:
Drug: Denosumab — Subcutaneous injection with 60 mg Denosumab once
  Other Names: Prolia
  Arms: Denosumab
Drug: Sodium chloride — Subcutaneous injection with NaCl once
  Other Names: NaCl
  Arms: Placebo

SUMMARY:
This RCT aims to assess whether treatment with Denosumab can improve semen quality in infertile men selected by serum AMH as a positive predictive biomarker.

DETAILED DESCRIPTION:
Background and rationale Infertility is a common problem globally and impaired semen quality is responsible for up to 40% of all cases. Despite the high prevalence there are currently only very limited treatment options to improve semen quality for infertile men. Instead, almost all infertile couples are treated with inseminations or assisted reproductive techniques (ARTs) independently of the etiology of infertility. ARTs are very successful but expensive and associated with a significant treatment burden of the female partner due to the invasive methodology and the need for hormonal treatment often for several months.

RANKL is a ligand for the receptor activator of nuclear factor κB (RANK), and their pathway plays a prominent role in the regulation of bone metabolism. The binding of RANKL to RANK on osteoclast precursors induces osteoclast maturation and activation, thereby stimulating bone resorption, and regulates cell cycle i.e., proliferation, differentiation, and apoptosis. Osteoprotegerin (OPG) is a secreted decoy receptor that controls RANKL-RANK interaction by binding RANKL and inhibits activation of RANK and preventing osteoclast differentiation and activation.

Denosumab, a drug used in millions of patients worldwide under trade names Prolia® and Xgeva®, inhibits the RANKL pathway and is used to treat osteoporosis and bone metastases. The drug's mechanism of action inhibits RANKL and thus inhibits bone resorption through reduced osteoclast activation. This reduces the loss of bone mineral density (BMD), which reduces the risk of bone loss and thereby the risk of fracture and osteoporosis. Denosumab has been shown in several clinical studies to be a safe and effective drug in both women and men and has been in clinical use in both sexes for many years. As Denosumab has a teratogenic effect, pharmacokinetic studies in both monkeys and healthy men were performed before approval of the drug as a treatment for osteoporosis in men. These studies showed that Denosumab concentration in semen does not pose a risk to the fetus during sexual intercourse with the pregnant woman and therefore is safe to use for the suggested infertility indication as there is no risk of fetal transmission.

Our research Recently, the research group has demonstrated the role of vitamin D in male reproduction by using functional animal studies supported by a randomized clinical trial. These investigations revealed that several bone factors such as Runx2, Osterix, FGF23, and in particular RANKL are expressed in the testis. The investigators found expression of RANKL in Sertoli cells, the receptor RANK in the testicular germ cells, and OPG in the peritubular cells in mice and human tissue. The presence of the RANKL system in these distinct testicular cell types indicates a possible direct effect on spermatogenesis.

The investigators therefore examined the effect of Denosumab in human testicular germ cell lines as well as in human testicular tissue ex vivo "hanging drop" cultures. Denosumab treatment in both cases increased the proliferation of the germinal cells. These studies confirmed that Denosumab treatment in vitro has a possibly beneficial effect on sperm production by reducing apoptosis in the germ cells. To further investigate this in vivo, the investigators injected the natural RANKL inhibitor OPG into mice daily for 14 days and compared them with their controls. Here, a a significantly increased testicular weight, increased thickness of germinal cell epithelium, and markedly higher sperm production was found. This prompted a human pilot study of 12 infertile men who besides infertility were healthy young men under 40 years of age. The men were treated with one 60 mg dosage of Denosumab subcutaneous (s.c.). The pilot study showed that as a group, the men's sperm production had increased 80 days after treatment. However, there was a large variation and 60% of men experienced an increase between 100-600% in sperm counts. The rest of the participants did not appear to benefit from the treatment. To validate putative biomarkers, a placebo controlled RCT was conducted in 100 infertile men with severe male infertility (Denosumab and Male Infertility: a RCT. ClinicalTrials.gov Identifier: NCT03030196). In this study, active treatment with 60 mg Denosumab s.c. was compared to placebo treatment. Importantly, there were no serious adverse reactions reported, nor severe hypocalcemia, nor abortions in the female partners of the patients. Data from this study has not been published yet.

In general, infertility in men is a heterogeneous disease but by identifying serum levels of AMH as a positive predictive biomarker, it seems the group of infertile men where treatment with Denosumab most likely will increase their semen quality can be selected.

Objective This RCT aims to assess whether treatment with Denosumab can improve semen quality in infertile men selected by serum AMH as a positive predictive biomarker.

Trial design and setting FITMI is a single-center, sponsor-investigator-initiated, placebo-controlled, double-blinded randomized clinical phase 2 trial. Following successful completion of screening procedures, subjects will be randomized in a 1:1 fashion to receive either Denosumab 60 mg s.c. or a placebo. The study will be carried out at the Department of Growth and Reproduction, Copenhagen University Hospital - Rigshospitalet, Copenhagen.

Analysis population Data will be analyzed using intention-to-treat (ITT) principles. When applying the ITT principle, all randomized participants will be analyzed in the groups to which the allocation originally was made, regardless of whether the participants received the intended treatment or whether a protocol violation or protocol deviation occurred. Participants who withdraw consent for the use of their data will not be included in any analysis and withdrawal of consent will be reported. A CONSORT flow diagram of participants will be presented in the study.

Sample size With the power to avoid a type II error set to 80% (1-β) at a two-sided 5% significance level 141 men in each of the investigation arms are needed to detect a difference in sperm concentration of 45% between intervention and placebo group in the primary outcome. A group-sequential design allows one interim analysis at half target recruitment. It is estimated that 1,300 infertile men will be screened as around 30% will meet the eligibility criteria and 70-75% will agree to participate in the trial. The calculations are based on the intra-individual variation in sperm concentration when including infertile men with sperm concentrations between 2 and 20 million pr. mL. It is expected that the placebo group will have a post-trial sperm concentration of 11 million pr. mL while the Denosumab group will have 16 million pr. mL with a maximum SD of 15. At an SD of 10, the same effect can be demonstrated by the inclusion of 170 men which is the basis for the interim analysis.

Statistics and underlying assumptions The primary analysis will be a covariance analysis in which day 80 measurements are regressed on baseline (including treatment assignment and subsequently AMH assignment). This will correctly take into account the grouped randomization scheme as well as the correlation between the day 80 and baseline measurements. Baseline is defined as the average of day -30 and 0 and Day 80 is defined as the average of day 80 and 83, unless abstinence time is <2 days or high fever which will result in exclusion of data. In both cases, data will be transformed as necessary to meet model assumptions. Subgroup analyses, e.g. for the group >9 mill/ml semen concentration will be performed. These analyses will not have the nominal type I error and will be interpreted as "hypothesis generating" results. Subsequently, subgroup analyses, e.g. for the group >9 mill/ml sperm concentration, low versus high baseline, FSH, Inhibin B and testis size and men with and without cryptorchidism and varicocele will be performed. Also, all regression analyses will be tested for major interactions between each covariate and the intervention variable. For each combination, it will be test whether the interaction term is significant and assess the effect size. When reporting a potentially relevant clinically significant effect, due diligence will be exercised because of the risk of type I errors when performing multiple tests.

Sperm concentration is subject to considerable intraindividual variation and a subgroup analysis will be performed in infertile men with less than 100% intraindividual variation to avoid a type 2 error

A predefined interim analysis described in detail in the protocol and in the publication of the study setup in Trials 2022 https://trialsjournal.biomedcentral.com/articles/10.1186/s13063-022-06478-4 will be performed after completion of 170 men.

ELIGIBILITY:
Inclusion Criterias:

* Infertile men ≥ 18 years and < 60 years of age
* Sperm concentration ≤ 20 million pr. mL
* Serum AMH levels ≥38 pmol/L.
* The participants must have appropriate Danish or English language skills and give written informed consent.

Exclusion Criterias:

* Chronic diseases, defined as diagnosis where signs, symptoms, and treatment imply an expected long duration and lack of a cure, such as diabetes mellitus, metabolism disorders, osteoporosis, colitis, etc.
* Sperm concentration <2 million pr. mL
* Men with current or previous malignancies, or at potential risk of testicular cancer after baseline examination and ultrasound will be excluded.
* Men with hypocalcemia at baseline, defined as ionized calcium of < 1,18 mmol/L or albumin corrected calcium < 2,17 mmol/L or total calcium < 2.14 mmol/L
* Serum vitamin D (25OHD) levels < 25 nmol/L
* eGFR < 60 mL/min/1,73 m2
* Insufficient dental status
* Vasectomy
* Semen volume < 0.9 mL
* Hypersensitivity to latex, Denosumab, or to any of the excipients (acetic acid, sodium hydroxide, Sorbitol (E420), Polysorbate 20) will be excluded.

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 180 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2024-10-22 (Actual); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
The difference in sperm concentration (million pr. mL) on day 80 | Day 80 and day 83 after inclusion
  Semen analysis - The average concentration of two semen samples delivered on day 80 and day 83 after inclusion is used.

SECONDARY OUTCOMES:
The difference in semen quality (total sperm count, motile sperm, progressive motile sperm and morphologically normal sperm) between baseline and two semen samples delivered at day 80 and day 83 after inclusion | Day 80 and day 83 after inclusion
  Semen analysis
The differences in pregnancies achieved spontaneously or by IUI before day 180 | Day 180 after inclusion
  Survey
The differences in live births where pregnancy is achieved spontaneously or at IUI before day 180 | Day 180 after inclusion
  Survey
The differences in number of live births where pregnancy is achieved by artificial insemination (IVF and ICSI) before day 180 | Day 180 after inclusion
  Survey
The difference in the number of miscarriages throughout the trial (IVF and ICSI) before day 180 | Day 450 after inclusion
  Survey
The difference in serum levels of FSH on day 80 | Day 80 after inclusion
  Serum sample
The difference in serum levels of reproductive hormone LH on day 80 | Day 80 after inclusion
  Serum sample
The difference in serum levels of reproductive hormone AMH on day 80 | Day 80 after inclusion
  Serum sample
The difference in serum levels of reproductive hormone Inhibin B on day 80 | Day 80 after inclusion
  Serum sample
The difference in serum levels of reproductive hormone SHBG on day 80 | Day 80 after inclusion
  Serum sample
The difference in serum levels of reproductive hormone INSL3 on day 80 | Day 80 after inclusion
  Serum sample
The difference in serum levels of reproductive hormone Testosterone on day 80 | Day 80 after inclusion
  Serum sample
The difference in serum levels of reproductive hormone estradiol on day 80 | Day 80 after inclusion
  Serum sample
The difference in gonadal function (Inhibin B/FSH ratio) on day 80 | Day 80 after inclusion
  Serum sample
The difference in gonadal function (Testosterone/LH ratio) on day 80 | Day 80 after inclusion
  Serum sample

OTHER OUTCOMES:
The change in testosterone/estradiol ratio on day 80 | Day 80 after inclusion
  Serum sample
The changes in serum levels of RANKL and OPG on day 80 | Day 80 after inclusion
  Serum sample
The changes in serum levels of OPG on day 80 | Day 80 after inclusion
  Serum sample
The changes in RANKL in seminal fluid on day 80 | Day 80 after inclusion
  Semen sample
The changes in OPG in seminal fluid on day 80 | Day 80 after inclusion
  Semen sample
The changes in AMH in seminal fluid on day 80 | Day 80 after inclusion
  Semen sample
The changes in Inhibin B in seminal fluid on day 80 | Day 80 after inclusion
  Semen sample
Changes of calcium in serum and seminal fluid on day 80 | Day 80 after inclusion
  Semen and serum sample
Changes of albumine in serum and seminal fluid on day 80 | Day 80 after inclusion
  Semen and serum sample
Changes of phosphate in serum and seminal fluid on day 80 | Day 80 after inclusion
  Semen and serum sample
Changes of magnesium in serum and seminal fluid on day 80 | Day 80 after inclusion
  Semen and serum sample
Changes of zinc in serum and seminal fluid on day 80 | Day 80 after inclusion
  Semen and serum sample
Changes of bicarbonate in serum and seminal fluid on day 80 | Day 80 after inclusion
  Semen and serum sample
Changes of citrate in serum and seminal fluid on day 80 | Day 80 after inclusion
  Semen and serum sample
Changes of PTH in serum and seminal fluid on day 80 | Day 80 after inclusion
  Semen and serum sample
Changes of VItamin D (25OHD) in serum and seminal fluid on day 80 | Day 80 after inclusion
  Semen and serum sample
Changes of creatinine (GFR) in serum and seminal fluid on day 80 | Day 80 after inclusion
  Semen and serum sample

CONTACTS AND LOCATIONS:
Overall Officials: Sam Kafai Yahyavi, MD, Principal Investigator — Rigshospitalet, Denmark; Rune Holt, MD, Principal Investigator — Rigshospitalet, Denmark
Locations (1):
- Department of Growth and Reproduction, Rigshospitalet, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Huynh T, Mollard R, Trounson A. Selected genetic factors associated with male infertility. Hum Reprod Update. 2002 Mar-Apr;8(2):183-98. doi: 10.1093/humupd/8.2.183. PMID 12099633
- [Background] Krausz C. Male infertility: pathogenesis and clinical diagnosis. Best Pract Res Clin Endocrinol Metab. 2011 Apr;25(2):271-85. doi: 10.1016/j.beem.2010.08.006. PMID 21397198
- [Background] Skakkebaek NE, Rajpert-De Meyts E, Buck Louis GM, Toppari J, Andersson AM, Eisenberg ML, Jensen TK, Jorgensen N, Swan SH, Sapra KJ, Ziebe S, Priskorn L, Juul A. Male Reproductive Disorders and Fertility Trends: Influences of Environment and Genetic Susceptibility. Physiol Rev. 2016 Jan;96(1):55-97. doi: 10.1152/physrev.00017.2015. PMID 26582516
- [Background] Blomberg Jensen M, Lawaetz JG, Petersen JH, Juul A, Jorgensen N. Effects of Vitamin D Supplementation on Semen Quality, Reproductive Hormones, and Live Birth Rate: A Randomized Clinical Trial. J Clin Endocrinol Metab. 2018 Mar 1;103(3):870-881. doi: 10.1210/jc.2017-01656. PMID 29126319
- [Background] Bollehuus Hansen L, Kaludjerovic J, Nielsen JE, Rehfeld A, Poulsen NN, Ide N, Skakkebaek NE, Frederiksen H, Juul A, Lanske B, Blomberg Jensen M. Influence of FGF23 and Klotho on male reproduction: Systemic vs direct effects. FASEB J. 2020 Sep;34(9):12436-12449. doi: 10.1096/fj.202000061RR. Epub 2020 Jul 30. PMID 32729975
- [Background] Juel Mortensen L, Lorenzen M, Jorgensen N, Andersson AM, Nielsen JE, Petersen LI, Lanske B, Juul A, Hansen JB, Blomberg Jensen M. Possible link between FSH and RANKL release from adipocytes in men with impaired gonadal function including Klinefelter syndrome. Bone. 2019 Jun;123:103-114. doi: 10.1016/j.bone.2019.03.022. Epub 2019 Mar 23. PMID 30914274
- [Background] Blomberg Jensen M. Vitamin D and male reproduction. Nat Rev Endocrinol. 2014 Mar;10(3):175-86. doi: 10.1038/nrendo.2013.262. Epub 2014 Jan 14. PMID 24419359
- [Background] Kearns AE, Khosla S, Kostenuik PJ. Receptor activator of nuclear factor kappaB ligand and osteoprotegerin regulation of bone remodeling in health and disease. Endocr Rev. 2008 Apr;29(2):155-92. doi: 10.1210/er.2007-0014. Epub 2007 Dec 5. PMID 18057140
- [Background] Lacey DL, Timms E, Tan HL, Kelley MJ, Dunstan CR, Burgess T, Elliott R, Colombero A, Elliott G, Scully S, Hsu H, Sullivan J, Hawkins N, Davy E, Capparelli C, Eli A, Qian YX, Kaufman S, Sarosi I, Shalhoub V, Senaldi G, Guo J, Delaney J, Boyle WJ. Osteoprotegerin ligand is a cytokine that regulates osteoclast differentiation and activation. Cell. 1998 Apr 17;93(2):165-76. doi: 10.1016/s0092-8674(00)81569-x. PMID 9568710
- [Background] Simonet WS, Lacey DL, Dunstan CR, Kelley M, Chang MS, Luthy R, Nguyen HQ, Wooden S, Bennett L, Boone T, Shimamoto G, DeRose M, Elliott R, Colombero A, Tan HL, Trail G, Sullivan J, Davy E, Bucay N, Renshaw-Gegg L, Hughes TM, Hill D, Pattison W, Campbell P, Sander S, Van G, Tarpley J, Derby P, Lee R, Boyle WJ. Osteoprotegerin: a novel secreted protein involved in the regulation of bone density. Cell. 1997 Apr 18;89(2):309-19. doi: 10.1016/s0092-8674(00)80209-3. PMID 9108485
- [Background] Khosla S. Minireview: the OPG/RANKL/RANK system. Endocrinology. 2001 Dec;142(12):5050-5. doi: 10.1210/endo.142.12.8536. PMID 11713196
- [Background] Anastasilakis AD, Toulis KA, Polyzos SA, Terpos E. RANKL inhibition for the management of patients with benign metabolic bone disorders. Expert Opin Investig Drugs. 2009 Aug;18(8):1085-102. doi: 10.1517/13543780903048929. PMID 19558335
- [Background] Makras P, Polyzos SA, Papatheodorou A, Kokkoris P, Chatzifotiadis D, Anastasilakis AD. Parathyroid hormone changes following denosumab treatment in postmenopausal osteoporosis. Clin Endocrinol (Oxf). 2013 Oct;79(4):499-503. doi: 10.1111/cen.12188. Epub 2013 Apr 1. PMID 23452098
- [Background] Schwarz P, Rasmussen AQ, Kvist TM, Andersen UB, Jorgensen NR. Paget's disease of the bone after treatment with Denosumab: a case report. Bone. 2012 May;50(5):1023-5. doi: 10.1016/j.bone.2012.01.020. PMID 22586699
- [Background] Polyzos SA, Singhellakis PN, Naot D, Adamidou F, Malandrinou FC, Anastasilakis AD, Polymerou V, Kita M. Denosumab treatment for juvenile Paget's disease: results from two adult patients with osteoprotegerin deficiency ("Balkan" mutation in the TNFRSF11B gene). J Clin Endocrinol Metab. 2014 Mar;99(3):703-7. doi: 10.1210/jc.2013-3762. Epub 2014 Jan 16. PMID 24433001
- [Background] Papapoulos S, Chapurlat R, Libanati C, Brandi ML, Brown JP, Czerwinski E, Krieg MA, Man Z, Mellstrom D, Radominski SC, Reginster JY, Resch H, Roman Ivorra JA, Roux C, Vittinghoff E, Austin M, Daizadeh N, Bradley MN, Grauer A, Cummings SR, Bone HG. Five years of denosumab exposure in women with postmenopausal osteoporosis: results from the first two years of the FREEDOM extension. J Bone Miner Res. 2012 Mar;27(3):694-701. doi: 10.1002/jbmr.1479. PMID 22113951
- [Background] Boonen S, Adachi JD, Man Z, Cummings SR, Lippuner K, Torring O, Gallagher JC, Farrerons J, Wang A, Franchimont N, San Martin J, Grauer A, McClung M. Treatment with denosumab reduces the incidence of new vertebral and hip fractures in postmenopausal women at high risk. J Clin Endocrinol Metab. 2011 Jun;96(6):1727-36. doi: 10.1210/jc.2010-2784. Epub 2011 Mar 16. PMID 21411557
- [Background] Sohn W, Lee E, Kankam MK, Egbuna O, Moffat G, Bussiere J, Padhi D, Ng E, Kumar S, Slatter JG. An open-label study in healthy men to evaluate the risk of seminal fluid transmission of denosumab to pregnant partners. Br J Clin Pharmacol. 2016 Feb;81(2):362-9. doi: 10.1111/bcp.12798. Epub 2015 Dec 5. PMID 26447647
- [Background] Bussiere JL, Pyrah I, Boyce R, Branstetter D, Loomis M, Andrews-Cleavenger D, Farman C, Elliott G, Chellman G. Reproductive toxicity of denosumab in cynomolgus monkeys. Reprod Toxicol. 2013 Dec;42:27-40. doi: 10.1016/j.reprotox.2013.07.018. Epub 2013 Jul 22. PMID 23886817
- [Background] Uhland AM, Kwiecinski GG, DeLuca HF. Normalization of serum calcium restores fertility in vitamin D-deficient male rats. J Nutr. 1992 Jun;122(6):1338-44. doi: 10.1093/jn/122.6.1338. PMID 1588451
- [Background] Kwiecinski GG, Petrie GI, DeLuca HF. Vitamin D is necessary for reproductive functions of the male rat. J Nutr. 1989 May;119(5):741-4. doi: 10.1093/jn/119.5.741. PMID 2723823
- [Background] Jorgensen A, Blomberg Jensen M, Nielsen JE, Juul A, Rajpert-De Meyts E. Influence of vitamin D on cisplatin sensitivity in testicular germ cell cancer-derived cell lines and in a NTera2 xenograft model. J Steroid Biochem Mol Biol. 2013 Jul;136:238-46. doi: 10.1016/j.jsbmb.2012.10.008. Epub 2012 Oct 23. PMID 23098692
- [Background] Blomberg Jensen M, Jorgensen A, Nielsen JE, Steinmeyer A, Leffers H, Juul A, Rajpert-De Meyts E. Vitamin D metabolism and effects on pluripotency genes and cell differentiation in testicular germ cell tumors in vitro and in vivo. Neoplasia. 2012 Oct;14(10):952-63. doi: 10.1593/neo.121164. PMID 23097629
- [Background] Blomberg Jensen M, Lieben L, Nielsen JE, Willems A, Jorgensen A, Juul A, Toppari J, Carmeliet G, Rajpert-De Meyts E. Characterization of the testicular, epididymal and endocrine phenotypes in the Leuven Vdr-deficient mouse model: targeting estrogen signalling. Mol Cell Endocrinol. 2013 Sep 5;377(1-2):93-102. doi: 10.1016/j.mce.2013.06.036. Epub 2013 Jul 11. PMID 23850520
- [Background] Blomberg Jensen M, Andreassen CH, Jorgensen A, Nielsen JE, Juel Mortensen L, Boisen IM, Schwarz P, Toppari J, Baron R, Lanske B, Juul A. RANKL regulates male reproductive function. Nat Commun. 2021 Apr 23;12(1):2450. doi: 10.1038/s41467-021-22734-8. PMID 33893301
- [Background] Adler RA, Gill RS. Clinical utility of denosumab for treatment of bone loss in men and women. Clin Interv Aging. 2011;6:119-24. doi: 10.2147/CIA.S14565. Epub 2011 May 24. PMID 21753866
- [Background] Boivin J, Bunting L, Collins JA, Nygren KG. International estimates of infertility prevalence and treatment-seeking: potential need and demand for infertility medical care. Hum Reprod. 2007 Jun;22(6):1506-12. doi: 10.1093/humrep/dem046. Epub 2007 Mar 21. PMID 17376819
- [Background] Lunenfeld B, Van Steirteghem A; Bertarelli Foundation. Infertility in the third millennium: implications for the individual, family and society: condensed meeting report from the Bertarelli Foundation's second global conference. Hum Reprod Update. 2004 Jul-Aug;10(4):317-26. doi: 10.1093/humupd/dmh028. Epub 2004 Jun 10. PMID 15192057
- [Derived] Yahyavi SK, Holt R, Jorsal MJ, Wall-Gremstrup G, Toft FB, Juel Mortensen L, Nohr B, Melsen LM, Praetorius L, Nielsen HS, Pinborg A, Beck Jensen JE, Schwarz P, Bennedbaek FN, Aksglaede L, Jorgensen A, Jorgensen N, Petersen JH, Juul A, Blomberg Jensen M. Effect of denosumab on semen quality in infertile men selected by serum level of antimullerian hormone: a randomized controlled trial. Fertil Steril. 2025 Oct;124(4):668-678. doi: 10.1016/j.fertnstert.2025.05.151. Epub 2025 May 20. PMID 40403914
- [Derived] Holt R, Yahyavi SK, Wall-Gremstrup G, Jorsal MJ, Toft FB, Jorgensen N, Juul A, Blomberg Jensen M. Low-serum antimullerian hormone is linked with poor semen quality in infertile men screened for participation in a randomized controlled trial. Fertil Steril. 2024 Aug;122(2):278-287. doi: 10.1016/j.fertnstert.2024.03.018. Epub 2024 Mar 24. PMID 38522503
- [Derived] Yahyavi SK, Holt R, Juel Mortensen L, Petersen JH, Jorgensen N, Juul A, Blomberg Jensen M. Effect of a single-dose denosumab on semen quality in infertile men (the FITMI study): study protocol for a randomized controlled trial. Trials. 2022 Jun 22;23(1):525. doi: 10.1186/s13063-022-06478-4. PMID 35733213